CLINICAL TRIAL: NCT04601558
Title: The Lifestyle Intervention on 10-year Year Risk of Cardiovascular Disease Among Women in the Form of Cochrane Abstracts: Randomized Controlled Trial
Brief Title: The Effect of Lifestyle Intervention on Cardiovascular Disease Risk Among Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: No. IP-2019-04-4882
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2020-10

CONDITIONS: Cardiovascular Risk Factor; Lifestyle Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): The first group of participants was control group. The number of participant was 70, and the participants in this group after recruitment received letter with their own cardiovascular risk factors and count of their 10-year risk of cardiovascular disease.
- Passive-intervention group (Sham Comparator): The second group of participant was passive-intervention group. There were 70 participants. This group of women after recruitment received letter with their own cardiovascular risk factors and count of their 10-year risk of cardiovascular disease. After this letter, every two months, they were receiving remainder on their own cardiovascular risk factors and count of their 10-year risk of cardiovascular disease.
  Interventions: Behavioral: The letters with remainder on cardiovascular risk factors
- Active-intervention group (Active Comparator): The third group of participant was active-intervention group. There were also 70 participants. This group of women after recruitment received letter with their own cardiovascular risk factors and count of their 10-year risk of cardiovascular disease. After this letter, every two months, active-intervention group were receiving Cochrane abstracts in the form of blog-shots.
  Interventions: Behavioral: The letters with the Cochrane abstracts in the form of blog-shots

INTERVENTIONS:
Behavioral: The letters with the Cochrane abstracts in the form of blog-shots — The active intervention were letters with the remainder on participant's own cardiovascular risk factors, a participant's own count of 10-year risk of cardiovascular disease, and Cochrane abstract in the form of blog-shots and personal advice in reducing cardiovascular disease risk.
  There were three Cochrane blog-shots. The first was about calcium in prevention of high blood pressure, the second was about the effect of reducing saturated fat acids in eating habits and the third consisted evidence of green and black tea for the prevention of cardiovascular diseases.
  The letters were sent three times, every two months after the participants received first letter about cardiovascular disease risk.
  Arms: Active-intervention group
Behavioral: The letters with remainder on cardiovascular risk factors — The passive intervention were letters with the remainder on participant's own cardiovascular risk factors and participant's own count of 10-year risk of cardiovascular disease.
  The letters were sent three times, every two months after the participants received first letter about cardiovascular disease risk.
  Arms: Passive-intervention group

SUMMARY:
Patient education in lifestyle changes has a positive effect on health in individuals with cardiovascular (CV) risk. Despite current positive evidence about lifestyle and dietary change in the prevention of CVD, the recommendations are still not consistently and optimally applied to women.

The aim of the study was to analyze the effect of an intervention in the form of Cochrane abstract letters on women between 45 to 65 years.

DETAILED DESCRIPTION:
The study took place in family medicine (FM) offices from 1 February 2018 to 1 June 2020. Two FM offices were in the city of Split, the capital of the Split-Dalmatian County, two offices were in Osijek, the capital of the Osijek-Baranja County, one in Kutina, and one in Rijeka.

The participants were all women between 45 to 65 years. The investigators enrolled 210 participants, and the participants were divided in three groups. The first group was control group, and participants were not exposed to the intervention. The second group was passive-intervention group, which means the participants received letters in the same time period as active-intervention group but only with a reminder at their own cardiovascular disease risk. The third group was active-intervention group, where the participants received letters every three months, with their own cardiovascular disease risk and Cochrane abstracts in the form of blog-shots.

The study participants first completed the Pre-study questionnaire (Questionnaire 1), which included: a) demographic data, b) attitudes and knowledge questionnaire about CV risk factors, c) decisional conflict scale (DCS), and d) integrative hope scale (IHS).

Attitudes and knowledge questionnaire about CV risk factors was created according to the model of "Ottawa Decision Support Tutorial".

The DCS consist of 16 items rated in a 5-point Likert-type response format, and measures individual's uncertainty toward a course of action. There are five subscales: uncertainty, informed, values clarity, support and effective decision. The scores on the total scale and subscales are calculated as a sum of items, divided by the number of items and multiplied by 25, allowing for a score range from zero (no decisional conflict) to 100 points (extreme decisional conflict). The Croatian version of the scale was previously validated.

The IHS is 23-items scale, a self-rating instrument with items being rated on a six-point Likert scale from 1, strongly disagree, to 6, strongly agree. It provides an overall score and four dimension scores, obtained by summing up the individual item scores, with negative items being rated inversely. This produces possible overall hope scores ranging from 23 to 138 with higher scores representing higher hopefulness. The scores for the sub-dimensions vary according to the number of items. The Croatian version of the scale was previously validated. Hope to be healthy at 70 and hope to reduce CV risk was assessed by a visual analogue scale from 0 to 100.

Ten-year risk of fatal CVD was estimated using the ACC/AHA (American College of Cardiology/American Heart Association) guidelines, based on the following data collected from the study participants: age, gender, race, total and HDL (high-density lipoprotein) cholesterol, systolic blood pressure, data about antihypertensive therapy, diabetes mellitus and smoking status. Also, BMI, waist and hip circumference, systolic and diastolic blood pressure, blood cholesterol, triglycerides, and smoking status were measured.

In the first months after recruitment, all participants received letter on home address with the count of their 10-year risk of cardiovascular disease.

After that, every two months, passive-intervention group and active-intervention group were receiving letters. The passive-intervention group of women were receiving the letters only with remainder on their own CV risk, and the active-intervention group were receiving Cochrane abstracts in the form of blog-shots.

There were three Cochrane blog-shots. The first was about calcium in prevention of high blood pressure, the second was about the effect of reducing saturated fat acids in eating habits and the third consisted informations of green and black tea for the prevention of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria

* female sex;
* age 45 to 65 years, with one or more CV risk factors [overweight or obesity, i. e. body mass index (BMI) ≥25 kg/m2, and/or central obesity - waist circumference ≥88 cm, high blood pressure (systolic blood pressure ≥140 mm Hg and/or diastolic blood pressure ≥90 mm Hg), high blood cholesterol (≥5.2 mmol/L) and active smoking];
* the participants on antihypertensive therapy were also included in the study.

Exclusion Criteria:

* current cardiovascular disease (ischemic heart disease, peripheral artery disease, and stroke) were excluded;
* the participants with malignant diseases;
* the participants with serious systemic disease;
* the participants with mental disease.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Ten-year Risk of Cardiovascular Disease (CVD) | Change from baseline 10-year risk of CVD at 6 months
  Ten-year risk of fatal CVD was estimated using the ACC/AHA (American College of Cardiology/American Heart Association) guidelines, based on the following data collected from the study participants: age, gender, race, total and HDL (high-density lipoprotein) cholesterol, systolic blood pressure, data about antihypertensive therapy, diabetes mellitus and smoking status.

SECONDARY OUTCOMES:
Weight | Change from baseline weight at 6 months
  Weight in kilograms (kg).
Body Mass Index (BMI) | Change from baseline BMI at 6 months
  Body mass index (BMI) is a person's weight in kilograms divided by the square of height in meters. A high BMI can be an indicator of high body fatness. BMI can be used to screen for weight categories that may lead to health problems but it is not diagnostic of the body fatness or health of an individual.
Waist Circumference | Change from baseline waist circumference at 6 months
  Waist circumference in centimeters (cm).
Hips Circumference | Change from baseline hips circumference at 6 months
  Hips circumference in centimeters (cm).
Smoking Status | Change from baseline smoking status at 6 months
  Smoking status related to continued or excessive smoking.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Split School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juric Petricevic S, Buljan I, Bjelanovic D, Mrduljas-Dujic N, Pekez T, Curkovic M, Vojvodic Z, Pavlicevic I, Marusic M, Marusic A. Effectiveness of letters to patients with or without Cochrane blogshots on 10-year cardiovascular risk change among women in menopausal transition: 6-month three-arm randomized controlled trial. BMC Med. 2022 Oct 20;20(1):381. doi: 10.1186/s12916-022-02555-2. PMID 36261832